CLINICAL TRIAL: NCT05506800
Title: Guangzhou Women's Health Cohort Study (GWHCS)
Status: Suspended | Type: Observational
Why Stopped: Due to the rebound of the COVID-19 epidemic in the city, we have to suspend the project temporarily.
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Head of the Department of Women's Health, Guangzhou Women and Children's Medical Center
Other Study IDs: 2021048B00
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Cervical Cancer; Breast Cancer; Lung Cancer; Colorectal Cancer; Endometrial Cancer; Ovarian Cancer; Hypertension; Diabetes; Reproductive Disorder
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Guangzhou Women's Health Cohort Study aims to explore the health trajectory and factors contributing to the health of women aged 35-64 in Guangzhou. Based on multiple population health registration data platforms, data of the cohort will provide information about the health of women across the lifespan, facilitating the decision-making process by local government . The cohort is progressing steadily, and the goal is to build a large women cohort covering 11 administrative districts of Guangzhou with a scale of 1 million by 2030.

DETAILED DESCRIPTION:
The Guangzhou Women's Health Cohort Study aims to explore the health trajectory and factors contributing to the health of women aged 35-64 in Guangzhou. Based on multiple population health registration data platforms, data of the cohort will provide information about the health of women across the lifespan, facilitating the decision-making process by local government . The cohort is progressing steadily, and the goal is to build a large women cohort covering 11 administrative districts of Guangzhou with a scale of 1 million by 2030.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 35-64 years old
* Women with registered permanent residence in Guangzhou
* Women with informed consent

Exclusion Criteria:

* Women without informed consent
* Women with reading and/or writing difficulties
* Women with serious mental disorders

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 35-64
Study Population: Women aged 35-64 years old with registered permanent residence in Guangzhou
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2016-03-03 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Incidence and mortality rate of cancer | through study completion, an average of 2 years
  Data from cancer registration platforms

SECONDARY OUTCOMES:
Hypertension and diabetes | through study completion, an average of 2 years
  Data from questionnaire
Reproductive health | through study completion, an average of 2 years
  Data from questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided